CLINICAL TRIAL: NCT05231304
Title: Retrospective Evaluation of Clinical and Radiographic Outcomes Following Total Talus Replacement
Acronym: RECLAIM
Status: Completed | Type: Observational
Sponsor: Restor3D (Industry)
Responsible Party: Sponsor
Other Study IDs: restor3d-002
Record Dates: First submitted 2022-01-27; First posted 2022-02-09 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Talus; Ankle Arthropathy
Keywords: Retrospective Study; Ankle Joint; Talus; Arthrodesis; Printing, Three-Dimensional; Joint Prosthesis; Prosthesis Design
MeSH Terms: conditions — Ankylosis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Total Talus Replacement
  Interventions: Procedure: Total Talus Replacement (TTR)
- Total Ankle Total Talus Replacement
  Interventions: Procedure: Total Ankle Total Talus Replacement (TATTR)
- Total Ankle Total Talus Replacement + Subtalar Fusion
  Interventions: Procedure: Total Ankle Total Talus Replacement + Subtalar Fusion (TATTR + STJ)
- Total Talus Replacement + Subtalar Fusion
  Interventions: Procedure: Total Talus Replacement + Subtalar Fusion (TTR + STJ)

INTERVENTIONS:
Procedure: Total Talus Replacement (TTR) — Surgical implantation of restor3d's patient-specific custom Total Talus Replacement device.
  Groups: Total Talus Replacement
Procedure: Total Ankle Total Talus Replacement (TATTR) — Surgical implantation of restor3d's patient-specific custom Total Ankle Total Talus Replacement (TATTR) device.
  Groups: Total Ankle Total Talus Replacement
Procedure: Total Ankle Total Talus Replacement + Subtalar Fusion (TATTR + STJ) — Surgical implantation of restor3d's patient-specific custom Total Ankle Total Talus Replacement (TATTR) device with concurrent subtalar fusion.
  Groups: Total Ankle Total Talus Replacement + Subtalar Fusion
Procedure: Total Talus Replacement + Subtalar Fusion (TTR + STJ) — Surgical implantation of restor3d's patient-specific custom Total Talus Replacement (TTR) device with concurrent subtalar fusion.
  Groups: Total Talus Replacement + Subtalar Fusion

SUMMARY:
This study is a retrospective analysis of patients who underwent surgery using a total talus replacement (TTR) implant with or without concurrent total ankle replacement and/or subtalar fusion. This study seeks to analyze the clinical and radiographic outcomes of TTR implant recipients and generate additional data on the safety and benefit of the TTR implant.

ELIGIBILITY:
Inclusion Criteria:

* >18 Years of Age
* Patient underwent surgery involving a total talus replacement implant between 1/1/2019 and 01/28/2022.

Exclusion Criteria:

* No available postoperative data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients who underwent surgery involving a TTR implant with or without total ankle replacement and/or subtalar fusion between 1/1/2019 and 01/28/2022 will be will be included in this retrospective review. Patients with at least one postoperative follow-up visit will be included in this study. Only data in existence as of 01/28/2022 will be collected.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2023-01-06 (Actual); Study Completion 2024-02-19 (Actual)

PRIMARY OUTCOMES:
Improvement in pain from pre-operative baseline | 12-months
  Primary probable benefit endpoint is improvement in pain at 12 months from preoperative baseline.

SECONDARY OUTCOMES:
Improvement in Patient Reported Outcomes | 3 months
  Secondary probably benefit endpoints will include patient reported functional outcome measures
Improvement in Patient Reported Outcomes | 6 months
  Secondary probably benefit endpoints will include patient reported functional outcome measures
Improvement in Patient Reported Outcomes | 12 months
  Secondary probably benefit endpoints will include patient reported functional outcome measures
Improvement in Patient Reported Outcomes | 24 months
  Secondary probably benefit endpoints will include patient reported functional outcome measures
Improvement in Patient Reported Outcomes | 36 months
  Secondary probably benefit endpoints will include patient reported functional outcome measures

OTHER OUTCOMES:
Subsequent Surgical Intervention | Up to 3 years.
  The primary safety outcome measure is rate of subsequent surgical intervention (SSI), as defined as any surgical procedure or service required after the initial implant of the TTR device.
Adverse Events (AEs)/Serious Adverse Events (SAEs) | Up to 3 years.
  Safety outcome measures by occurrence of adverse events (AEs), device- or procedure related AEs, and serious AEs.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Orthopaedic Institute of Western Kentucky, Paducah, Kentucky
  - The Bellevue Hospital, Bellevue, Ohio